CLINICAL TRIAL: NCT05008393
Title: Efficacy of PJS-539 for Adult Patients With SARS-CoV-2: Multicentre, Phase 2, Randomized, Double-blind, Placebo-controlled Clinical Trial.
Brief Title: Efficacy of PJS-539 for Adult Patients With COVID-19.
Acronym: PJS-539
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital do Coracao (Other)
Collaborators: Covicept (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IP-HCOR/PJS-539; Phase2_PJS-539 (Other: IP-HCor)
Record Dates: First submitted 2021-08-16; First posted 2021-08-17 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-02

CONDITIONS: Covid19; COVID-19 Pneumonia
Keywords: COVID-19; Antiviral
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Patients will be randomized at a 1: 1: 1 ratio to each of the treatment groups.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The placebo used in this study will consist of the diluent solution used in the interventional drug preparation, which has the same physical characteristics as the interventional drug preparation. All the solutions will be prepared at a central pharmacy and will be sent to each site center in specific boxes containing the necessary regulatory information. The solutions for each study arm will be identified by a random letter from A to I (three letters each arm).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Patients will receive placebo orally once daily for 10 days.
  Interventions: Drug: Placebo
- PJS-539 Dose 1 (Experimental): Patients will receive PJS-539 dose 1 orally once daily for 10 days.
  Interventions: Drug: PJS-539 Dose 1
- PJS-539 Dose 2 (Experimental): Patients will receive PJS-539 dose 2 orally once daily for 10 days.
  Interventions: Drug: PJS-539 Dose 2

INTERVENTIONS:
Drug: PJS-539 Dose 1 — Patients will receive PJS-539 dose 1 daily for 10 days.
  Arms: PJS-539 Dose 1
Drug: PJS-539 Dose 2 — Patients will receive PJS-539 Dose 2 daily for 10 days.
  Arms: PJS-539 Dose 2
Drug: Placebo — Patients will receive placebo daily for 10 days.
  Arms: Placebo

SUMMARY:
The PJS-539 is a multicentre, phase 2, randomized, double-blind, placebo-controlled clinical trial to evaluate the effect of PJS-539 in the viral load of patients with severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2).

DETAILED DESCRIPTION:
COVID-19, a disease caused by severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) became a pandemic in March 2020. Clinically, the coronavirus disease 2019 (COVID-19) ranges from asymptomatic disease in some to severe forms. However, until now, only the use of corticosteroids in selected patients has been shown to improve clinical outcomes in patients with COVID-19.

PJS-539 has been demonstrated to inhibit viral uptake and replication of SARS-CoV-2.

The objective of this Phase II trial is to assess the effect of PJS-539 in the viral load of patients with mild to moderate COVID-19 symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (age ≥ 18 years);
2. COVID-19 diagnosis confirmed by:

   1. Detection of SARS-CoV-2 by reverse transcription polymerase chain reaction (RT-PCR), or
   2. Rapid genetic or antigen tests validated by Brazilian National Health Surveillance Agency (ANVISA);
3. Mild or moderate symptoms without indication for hospitalization;
4. Symptoms started seven days ago or less;
5. Be able to access the study's online questionnaire.

Exclusion Criteria:

1. Pregnant or lactating women;
2. Known allergy or hypersensitivity to the study drug;
3. Patients at high risk of bleeding, defined by:

   1. Previous Intracranial hemorrhage,
   2. Ischemic stroke in the last 3 months,
   3. Anatomical vascular alteration of the central nervous system known, such as aneurysms or arteriovenous malformations,
   4. Malignant neoplasm of the central nervous system known,
   5. Metastatic solid neoplasia,
   6. Significant closed head or facial trauma in the last 3 months (defined as any trauma that required medical evaluation or hospitalization),
   7. Known intracranial abnormalities not listed as absolute contraindications (e.g., benign intracranial tumor),
   8. Bleeding in the last 2 to 4 weeks (excluding menstrual bleeding),
   9. Surgical procedure in the last 3 weeks,
   10. Current use of full-dose anticoagulants (warfarin, enoxaparin or new anticoagulants) or dual antiplatelet therapy,
   11. Thrombocytopenia (<100,000/mL) or international normalized ratio (INR) > 1.3;
4. Renal failure, defined as glomerular filtration rate (GFR) estimated by the formulas Modification of Diet in Renal Disease (MDRD) or Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) <30 mL/min/1.73m2;
5. Previous participation in the study;
6. History of liver disease (cirrhosis) reported by the patient or in medical records, presence of esophageal varices or presence of ascites;
7. Decompensated heart failure, defined by the presence of dyspnea attributed to cardiac cause, edema of the lower limbs, crackles on pulmonary auscultation or pathological jugular turgency.
8. Participation in other clinical trials with antivirals in COVID-19

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2021-09-25 (Actual); Primary Completion 2022-02-03 (Actual); Study Completion 2022-03-04 (Actual)

PRIMARY OUTCOMES:
Decay rate of the SARS-CoV-2 viral load. | At day 10
  Decay rate of the SARS-CoV-2 viral load logarithmic curve obtained via nasopharyngeal swab between the baseline and the fifth and tenth days after randomization.

SECONDARY OUTCOMES:
Hospital admission | Day 28
  Need for hospital admission.
Need for invasive mechanical ventilation | Day 28
  Intubation and initiation of mechanical ventilation for any given reason
Time to symptoms resolution | Day 10
  Time from randomization to symptoms resolution
Ordinal clinical scale of symptoms | Day 14
  Evaluation of the clinical scale of symptoms, which ranges from 1 to 7 as follows: 1. not hospitalized, without limitation of daily activities; 2. not hospitalized, with limitation of daily activities; 3. hospitalized, without the need for supplemental oxygen; 4. hospitalized, requiring supplemental oxygen; 5 hospitalized, requiring high-flow nasal oxygen therapy, non-invasive mechanical ventilation, or both; 6. hospitalized, requiring blood oxygenation through a membrane system, invasive mechanical ventilation, or both; 7. Death.
Adverse events | Up to 28 days
  Grade 1, 2, 3 and 4 adverse events, which were not present at the patient's entrance, defined by the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events
Bleeding | Up to 28 days
  Defines as:
  Major: Defined as clinical bleeding associated with any of the following: fatal outcome, critical site involvement (intracranial, intraspinal, intraocular, pericardial, intra-articular, intramuscular with compartmental or retroperitoneal syndrome), or clinical bleeding with a drop in hemoglobin concentration ≥2g/dL, or need for transfusion of ≥2 units of packed red blood cells or whole blood. All intracerebral (or intraparenchymal) bleeds are included in the primary analysis as hemorrhagic stroke.
  Clinically relevant non-major: Defined as clinical bleeding that does not present major bleeding criteria, but requires medical intervention, unscheduled contact (in person or by telephone) with a doctor, temporary interruption of the study drug, pain or impairment of daily activities.
  Minor: Defined as clinical bleeding that does not meet criteria for clinically relevant major or non-major bleeding.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Tomazini, MD, Principal Investigator — Hospital do Coracao; Alexandre Biasi Cavalcanti, MD, PhD, Study Director — Hospital do Coracao
Locations (1):
- Hospital do Coracao, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No